CLINICAL TRIAL: NCT01818063
Title: An Adaptive, Randomized Phase II Trial to Determine Pathologic Complete Response With the Addition of Carboplatin With and Without Veliparib to Standard Chemotherapy in the Neoadjuvant Treatment of Triple-Negative Breast Cancer
Brief Title: Carboplatin and Combination Chemotherapy With or Without Veliparib in Treating Patients With Stage IIB-IIIC Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12G.376; 2012-47 (Other: CCRRC); JT 2997 (Other: JeffTrial Number)
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Doxorubicin; liposomal doxorubicin; Cyclophosphamide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel IV and carboplatin IV on day 1 (course 1 only) or day 2 (courses 2-12). Treatment repeats every 7 days for 12 courses in the absence of disease progression or unacceptable toxicity. Beginning 21 days after the last course, patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm 2 (veliparib, paclitaxel, carboplatin) (Experimental): Patients receive veliparib PO BID on days 1-5. Patients also receive paclitaxel IV and carboplatin IV on day 3 (course 1 only) or day 4 (courses 2-12). Treatment repeats every 7 days for 12 courses in the absence of disease progression or unacceptable toxicity. Beginning 21 days after the last course, patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Veliparib

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Taxol; Abraxane
Drug: Carboplatin — Given IV
  Other Names: cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II); Paraplatin; Paraplatin-AQ
Drug: Doxorubicin — Given IV
  Other Names: Adriamycin; hydroxydaunorubicin; Adriamycin PFS; Adriamycin RDF; Rubex; Doxil
Drug: Cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane; Lyophilizedcytoxan
Drug: Veliparib — Given PO
  Other Names: ABT-888
  Arms: Arm 2 (veliparib, paclitaxel, carboplatin)

SUMMARY:
This randomized phase II trial studies how well carboplatin and combination chemotherapy with or without veliparib works in treating patients with stage IIB-IIIC breast cancer. Drugs used in chemotherapy, such as paclitaxel, carboplatin, doxorubicin hydrochloride, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving carboplatin and combination chemotherapy are more effective with or without veliparib is more effective in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1) To compare the pathologic complete response (path CR) in patients with stage IIB or stage III triple negative breast cancer treated with neoadjuvant paclitaxel and carboplatin to the path CR of patients treated with paclitaxel, carboplatin, and veliparib.

SECONDARY OBJECTIVES:

1. Relapse free survival (follow-up period of 36 months).
2. Overall clinical response to neoadjuvant therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) and carboplatin IV on day 1 (course 1 only) or day 2 (courses 2-12). Treatment repeats every 7 days for 12 courses in the absence of disease progression or unacceptable toxicity. Beginning 21 days after the last course, patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive veliparib orally (PO) twice daily (BID) on days 1-5. Patients also receive paclitaxel IV and carboplatin IV on day 3 (course 1 only) or day 4 (courses 2-12). Treatment repeats every 7 days for 12 courses in the absence of disease progression or unacceptable toxicity. Beginning 21 days after the last course, patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any study-related procedures.
2. Histologically confirmed adenocarcinoma of the breast with the following markers: Estrogen receptor negative (<1%), progesterone receptor negative (<1%), and Her-2/neu negative (Her-2/neu 0-1+ IHC or FISH ratio <1.8 or average HER2 gene copy number of <four signal/nucleus for test systems without internal control probe).
3. Female ≥ 18 years old.
4. Clinical stage IIA (T2N0), IIB (T2N1, T3N0) or stage IIIA (T1N2, T2N2, T3N1, T3N2), IIIB, or IIIC breast cancer with no prior treatment.
5. Complete radiology or tumor assessment within 28 days prior to enrollment

   1. Breast MRI
   2. Unilateral Breast Ultrasound
   3. Distant metastatic work-up completed with PET/CT.
   4. If enlarged axillary lymph nodes are found during staging scans, FNA must be performed to determine whether the node is involved with cancer.
   5. If axillary lymph nodes are clinically negative during initial work-up, sentinel node biopsy will be performed prior to initiation of chemotherapy.
6. ECOG Performance Status of 0 or 1
7. Adequate organ and hematologic function as evidenced by the following laboratory studies within 4 weeks of study enrollment:

   1. Cardiac Ejection Fraction >/= lower limit of normal as determined by 2-D echo or MUGA scan according to institutional standards.
   2. Hematologic function, as follows: Absolute neutrophil count ≥ 1.5 x 109/L, Platelet count ≥ 100 x 109/L and ≤ 850 x 109/L, Hemoglobin ≥ 9 g/dL, PTT and INR < 1.5 x ULN.
   3. Renal function, as follows: Serum creatinine </= 1.4 mg/dL).
   4. Hepatic function, as follows:Aspartate aminotransferase (AST) ≤ 2.5 x ULN, Alanine aminotransferase (ALT) ≤ 2.5 x ULN , Total bilirubin ≤ 2 x ULN (except for patients with UGT1A1 promoter polymorphism, i.e. Gilbert syndrome, confirmed by genotyping or Invader UGT1A1 molecular assay prior to study enrollment. Patients enrolled with Gilbert syndrome must have total bilirubin < 3 ULN).
8. Patient must be willing and able to undergo MRI as outlined in protocol.

Exclusion Criteria:

1. Known hypersensitivity to doxorubicin, cyclophosphamide, paclitaxel, cremophor or medications containing cremophor(miconazole, docetaxel, sandimmune, nelfinavir mesylate, propofol, diazepam injection, vitamin K injection, ixabepilone, aci-jel) or carboplatin.
2. Known HIV or active Hepatitis B or C infection.
3. Prior treatment for the currently diagnosed breast cancer.
4. Prior treatment with doxorubicin up to 400 mg/m2.
5. Pre-existing Grade 3 or 4 sensory neuropathy.
6. History of bleeding diathesis or extensive bleeding requiring blood transfusion within 14 days of enrollment.
7. Major surgical procedure within 4 weeks (28 days) prior to enrollment (port placement is not considered a major surgical procedure).
8. Clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, congestive heart failure, or ongoing arrhythmias requiring medication or pacemaker.
9. Non-healing wound, ulcer or fracture.
10. Ongoing or active infection.
11. Pregnant (i.e., positive beta-human chorionic gonadotropin test) or lactating
12. Not willing to use a highly effective method of birth control (i.e. those which result in low failure rates, less than 1% per year), defined as intrauterine devices, barrier methods (condoms, contraceptive sponges, diaphragms, vaginal rings used with spermicidal jellies or creams), oral contraceptive pills, or sexual abstinence. Contraception must be used during the study.
13. T0 tumors
14. Active dental infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Mitchell, MD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania

REFERENCES:
- [Background] Perou CM. Molecular stratification of triple-negative breast cancers. Oncologist. 2011;16 Suppl 1:61-70. doi: 10.1634/theoncologist.2011-S1-61. PMID 21278442
- [Background] Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4429-34. doi: 10.1158/1078-0432.CCR-06-3045. PMID 17671126
- [Background] Bauer KR, Brown M, Cress RD, Parise CA, Caggiano V. Descriptive analysis of estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and HER2-negative invasive breast cancer, the so-called triple-negative phenotype: a population-based study from the California cancer Registry. Cancer. 2007 May 1;109(9):1721-8. doi: 10.1002/cncr.22618. PMID 17387718
- [Background] Lund MJ, Butler EN, Bumpers HL, Okoli J, Rizzo M, Hatchett N, Green VL, Brawley OW, Oprea-Ilies GM, Gabram SG. High prevalence of triple-negative tumors in an urban cancer center. Cancer. 2008 Aug 1;113(3):608-15. doi: 10.1002/cncr.23569. PMID 18484596
- [Background] Bosch A, Eroles P, Zaragoza R, Vina JR, Lluch A. Triple-negative breast cancer: molecular features, pathogenesis, treatment and current lines of research. Cancer Treat Rev. 2010 May;36(3):206-15. doi: 10.1016/j.ctrv.2009.12.002. Epub 2010 Jan 8. PMID 20060649
- [Background] NCCN. NCCN Clinical Practice Guidelines in Oncology, Version 2.2011. 2011.
- [Background] Henderson IC, Berry DA, Demetri GD, Cirrincione CT, Goldstein LJ, Martino S, Ingle JN, Cooper MR, Hayes DF, Tkaczuk KH, Fleming G, Holland JF, Duggan DB, Carpenter JT, Frei E 3rd, Schilsky RL, Wood WC, Muss HB, Norton L. Improved outcomes from adding sequential Paclitaxel but not from escalating Doxorubicin dose in an adjuvant chemotherapy regimen for patients with node-positive primary breast cancer. J Clin Oncol. 2003 Mar 15;21(6):976-83. doi: 10.1200/JCO.2003.02.063. PMID 12637460
- [Background] Mamounas EP, Bryant J, Lembersky B, Fehrenbacher L, Sedlacek SM, Fisher B, Wickerham DL, Yothers G, Soran A, Wolmark N. Paclitaxel after doxorubicin plus cyclophosphamide as adjuvant chemotherapy for node-positive breast cancer: results from NSABP B-28. J Clin Oncol. 2005 Jun 1;23(16):3686-96. doi: 10.1200/JCO.2005.10.517. Epub 2005 May 16. PMID 15897552
- [Background] Sparano JA, Wang M, Martino S, Jones V, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Weekly paclitaxel in the adjuvant treatment of breast cancer. N Engl J Med. 2008 Apr 17;358(16):1663-71. doi: 10.1056/NEJMoa0707056. PMID 18420499
- [Background] Liedtke C, Mazouni C, Hess KR, Andre F, Tordai A, Mejia JA, Symmans WF, Gonzalez-Angulo AM, Hennessy B, Green M, Cristofanilli M, Hortobagyi GN, Pusztai L. Response to neoadjuvant therapy and long-term survival in patients with triple-negative breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1275-81. doi: 10.1200/JCO.2007.14.4147. Epub 2008 Feb 4. PMID 18250347
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903
- [Background] Wang S, Yang H, Tong F, Zhang J, Yang D, Liu H, Cao Y, Liu P, Zhou P, Cheng L, Liu M, Guo J. Response to neoadjuvant therapy and disease free survival in patients with triple-negative breast cancer. Gan To Kagaku Ryoho. 2009 Feb;36(2):255-8. PMID 19223741
- [Background] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Background] Perez EA, Moreno-Aspitia A, Aubrey Thompson E, Andorfer CA. Adjuvant therapy of triple negative breast cancer. Breast Cancer Res Treat. 2010 Apr;120(2):285-91. doi: 10.1007/s10549-010-0736-z. Epub 2010 Jan 22. PMID 20094772
- [Background] Sirohi B, Arnedos M, Popat S, Ashley S, Nerurkar A, Walsh G, Johnston S, Smith IE. Platinum-based chemotherapy in triple-negative breast cancer. Ann Oncol. 2008 Nov;19(11):1847-52. doi: 10.1093/annonc/mdn395. Epub 2008 Jun 20. PMID 18567607
- [Background] Roy V, Pockaj BA, Allred JB, Apsey H, Northfelt DW, Nikcevich D, Mattar B, Perez EA. A Phase II trial of docetaxel and carboplatin administered every 2 weeks as preoperative therapy for stage II or III breast cancer: NCCTG study N0338. Am J Clin Oncol. 2013 Dec;36(6):540-4. doi: 10.1097/COC.0b013e318256f619. PMID 22868240
- [Background] Frasci G, Comella P, Rinaldo M, Iodice G, Di Bonito M, D'Aiuto M, Petrillo A, Lastoria S, Siani C, Comella G, D'Aiuto G. Preoperative weekly cisplatin-epirubicin-paclitaxel with G-CSF support in triple-negative large operable breast cancer. Ann Oncol. 2009 Jul;20(7):1185-92. doi: 10.1093/annonc/mdn748. Epub 2009 Feb 13. PMID 19218307
- [Background] Anders CK, Winer EP, Ford JM, Dent R, Silver DP, Sledge GW, Carey LA. Poly(ADP-Ribose) polymerase inhibition: "targeted" therapy for triple-negative breast cancer. Clin Cancer Res. 2010 Oct 1;16(19):4702-10. doi: 10.1158/1078-0432.CCR-10-0939. Epub 2010 Sep 21. PMID 20858840
- [Background] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- [Background] O'Shaughnessy J, Osborne C, Pippen JE, Yoffe M, Patt D, Rocha C, Koo IC, Sherman BM, Bradley C. Iniparib plus chemotherapy in metastatic triple-negative breast cancer. N Engl J Med. 2011 Jan 20;364(3):205-14. doi: 10.1056/NEJMoa1011418. Epub 2011 Jan 5. PMID 21208101
- [Background] O'Shaughnessy J, Schwartzberg S, Danso M, Rugo H, Miller K, Yardley D. A randomized phase III study of iniparib (BSI-201) in combination with gemcitabine/carboplatin (G/C) in metastatic triple-negative breast cancer (TNBC). J Clin Oncol 2011;29 (suppl; abstr 1007).
- [Background] Liu X, Shi Y, Maag DX, Palma JP, Patterson MJ, Ellis PA, Surber BW, Ready DB, Soni NB, Ladror US, Xu AJ, Iyer R, Harlan JE, Solomon LR, Donawho CK, Penning TD, Johnson EF, Shoemaker AR. Iniparib nonselectively modifies cysteine-containing proteins in tumor cells and is not a bona fide PARP inhibitor. Clin Cancer Res. 2012 Jan 15;18(2):510-23. doi: 10.1158/1078-0432.CCR-11-1973. Epub 2011 Nov 29. PMID 22128301
- [Background] Patel AG, De Lorenzo SB, Flatten KS, Poirier GG, Kaufmann SH. Failure of iniparib to inhibit poly(ADP-Ribose) polymerase in vitro. Clin Cancer Res. 2012 Mar 15;18(6):1655-62. doi: 10.1158/1078-0432.CCR-11-2890. Epub 2012 Jan 30. PMID 22291137
- [Background] Comen EA, Robson M. Poly(ADP-ribose) polymerase inhibitors in triple-negative breast cancer. Cancer J. 2010 Jan-Feb;16(1):48-52. doi: 10.1097/PPO.0b013e3181cf01eb. PMID 20164690
- [Background] Chen XS, Nie XQ, Chen CM, Wu JY, Wu J, Lu JS, Shao ZM, Shen ZZ, Shen KW. Weekly paclitaxel plus carboplatin is an effective nonanthracycline-containing regimen as neoadjuvant chemotherapy for breast cancer. Ann Oncol. 2010 May;21(5):961-7. doi: 10.1093/annonc/mdq041. Epub 2010 Mar 8. PMID 20211870
- [Background] Betensky RA, Louis DN, Cairncross JG. Influence of unrecognized molecular heterogeneity on randomized clinical trials. J Clin Oncol. 2002 May 15;20(10):2495-9. doi: 10.1200/JCO.2002.06.140. PMID 12011127
- [Background] Berry DA. Bayesian clinical trials. Nat Rev Drug Discov. 2006 Jan;5(1):27-36. doi: 10.1038/nrd1927. PMID 16485344
- [Background] Barker AD, Sigman CC, Kelloff GJ, Hylton NM, Berry DA, Esserman LJ. I-SPY 2: an adaptive breast cancer trial design in the setting of neoadjuvant chemotherapy. Clin Pharmacol Ther. 2009 Jul;86(1):97-100. doi: 10.1038/clpt.2009.68. Epub 2009 May 13. PMID 19440188
- [Background] Heagerty PJ, Zheng Y. Survival model predictive accuracy and ROC curves. Biometrics. 2005 Mar;61(1):92-105. doi: 10.1111/j.0006-341X.2005.030814.x. PMID 15737082
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Background] Chen JQ, Russo J. ERalpha-negative and triple negative breast cancer: molecular features and potential therapeutic approaches. Biochim Biophys Acta. 2009 Dec;1796(2):162-75. doi: 10.1016/j.bbcan.2009.06.003. Epub 2009 Jun 13. PMID 19527773
- [Background] Hergueta-Redondo M, Palacios J, Cano A, Moreno-Bueno G. "New" molecular taxonomy in breast cancer. Clin Transl Oncol. 2008 Dec;10(12):777-85. doi: 10.1007/s12094-008-0290-x. PMID 19068448
- [Background] Rakha EA, Reis-Filho JS, Ellis IO. Basal-like breast cancer: a critical review. J Clin Oncol. 2008 May 20;26(15):2568-81. doi: 10.1200/JCO.2007.13.1748. PMID 18487574
- [Background] Holstege H, Joosse SA, van Oostrom CT, Nederlof PM, de Vries A, Jonkers J. High incidence of protein-truncating TP53 mutations in BRCA1-related breast cancer. Cancer Res. 2009 Apr 15;69(8):3625-33. doi: 10.1158/0008-5472.CAN-08-3426. Epub 2009 Mar 31. PMID 19336573
- [Background] Lakhani SR, Reis-Filho JS, Fulford L, Penault-Llorca F, van der Vijver M, Parry S, Bishop T, Benitez J, Rivas C, Bignon YJ, Chang-Claude J, Hamann U, Cornelisse CJ, Devilee P, Beckmann MW, Nestle-Kramling C, Daly PA, Haites N, Varley J, Lalloo F, Evans G, Maugard C, Meijers-Heijboer H, Klijn JG, Olah E, Gusterson BA, Pilotti S, Radice P, Scherneck S, Sobol H, Jacquemier J, Wagner T, Peto J, Stratton MR, McGuffog L, Easton DF; Breast Cancer Linkage Consortium. Prediction of BRCA1 status in patients with breast cancer using estrogen receptor and basal phenotype. Clin Cancer Res. 2005 Jul 15;11(14):5175-80. doi: 10.1158/1078-0432.CCR-04-2424. PMID 16033833
- [Background] Thiery JP, Acloque H, Huang RY, Nieto MA. Epithelial-mesenchymal transitions in development and disease. Cell. 2009 Nov 25;139(5):871-90. doi: 10.1016/j.cell.2009.11.007. PMID 19945376
- [Background] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166
- [Background] Ruckhaberle E, Karn T, Engels K, Turley H, Hanker L, Muller V, Schmidt M, Ahr A, Gaetje R, Holtrich U, Kaufmann M, Rody A. Prognostic impact of thymidine phosphorylase expression in breast cancer--comparison of microarray and immunohistochemical data. Eur J Cancer. 2010 Feb;46(3):549-57. doi: 10.1016/j.ejca.2009.11.020. Epub 2009 Dec 18. PMID 20022486
- [Background] Palacios J, Honrado E, Osorio A, Cazorla A, Sarrio D, Barroso A, Rodriguez S, Cigudosa JC, Diez O, Alonso C, Lerma E, Dopazo J, Rivas C, Benitez J. Phenotypic characterization of BRCA1 and BRCA2 tumors based in a tissue microarray study with 37 immunohistochemical markers. Breast Cancer Res Treat. 2005 Mar;90(1):5-14. doi: 10.1007/s10549-004-1536-0. PMID 15770521
- [Background] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer. Arch Pathol Lab Med. 2010 Jun;134(6):907-22. doi: 10.5858/134.6.907. PMID 20524868
- [Background] Vance GH, Barry TS, Bloom KJ, Fitzgibbons PL, Hicks DG, Jenkins RB, Persons DL, Tubbs RR, Hammond ME; College of American Pathologists. Genetic heterogeneity in HER2 testing in breast cancer: panel summary and guidelines. Arch Pathol Lab Med. 2009 Apr;133(4):611-2. doi: 10.5858/133.4.611. PMID 19391661
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants That Achieve Pathologic Complete Response (PCR)
Description: PCR is defined as the absence of any residual invasive cancer on hematoxylin and eosin (H&E) evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes.
Time Frame: 36 months following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 5 | 4
Participants | 3 | 3

2. Secondary Outcome: Overall Clinical Response
Description: The count and percentage of subjects with each category of overall clinical response will be summarized by presence of baseline measureable disease (i.e., complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD], unable to evaluate [UE], neurogenerative disease [ND]). Evaluated per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) as assessed b MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  Beta will be used as priors for combination regimens in calculating the posterior distribution of the pathologic complete response [pCR] for each respective treatment group. Among subjects with measurable disease, a 95% credible region will be calculated for the odds ratio for each treatment combination relative to each other.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 5 | 4
Participants
  Progressive Disease | 1 | 1
  Partial Response | 2 | 1
  Pathological Complete Response | 2 | 2

3. Secondary Outcome: Relapse Free Survival
Description: Analyzed using Kaplan-Meier methods, stratified by study group, and the log rank test will be completed.
Time Frame: Up to 3 years
Population: Sincere efforts have been made to gather and report the data, however, no data is available for this outcome measure.
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 (Paclitaxel, Carboplatin) | Arm 2 (Veliparib, Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Paclitaxel, Carboplatin) (N=5) | Arm 2 (Veliparib, Paclitaxel, Carboplatin) (N=4)
Viral Meningitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Paclitaxel, Carboplatin) (N=5) | Arm 2 (Veliparib, Paclitaxel, Carboplatin) (N=4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Alkaline phosphatase Increased (Blood and lymphatic system disorders) | 1 (7) | 1 (1)
ALT Increase (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bone Pain (General disorders) | 2 (7) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dehydration (General disorders) | 1 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (3) | 1 (2)
Head Injury (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Hot flashes (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Infection UTI (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 1 (2)
Laryngeal Inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Night Sweats (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Platelet Count decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Psychiatric Disorders, mood (Psychiatric disorders) | 0 (0) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Runny nose (General disorders) | 0 (0) | 1 (1)
Scalp pain (General disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Scratch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Voice alteration (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes